CLINICAL TRIAL: NCT06218732
Title: Understanding Participation Habits: An Observational Investigation Within Semantic Dementia Clinical Trials
Brief Title: Revealing Engagement Dynamics Among Semantic Dementia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 58672364
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Semantic Dementia
Keywords: Semantic Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study intends to investigate the personal experiences of semantic dementia patients who take part in a separate clinical study including a specific medication intervention. The major focus will be on closely following individuals' rates of trial completion and withdrawal.

The data collected from this study will help improve future outcomes for all semantic dementia as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with semantic dementia
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with semantic dementia who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a semantic dementia clinical research. | 3 months
Number of semantic dementia study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paplikar A, Vandana VP, Mekala S, Darshini KJ, Arshad F, Iyer GK, Kandukuri R, Divyaraj G, Varghese F, Kaul S, Patterson K, Alladi S. Semantic memory impairment in dementia: A cross-cultural adaptation study. Neurol Sci. 2022 Jan;43(1):265-273. doi: 10.1007/s10072-021-05272-5. Epub 2021 May 8. PMID 33966130
- [Background] Kertesz A, Jesso S, Harciarek M, Blair M, McMonagle P. What is semantic dementia?: a cohort study of diagnostic features and clinical boundaries. Arch Neurol. 2010 Apr;67(4):483-9. doi: 10.1001/archneurol.2010.55. PMID 20385916
- [Background] Sato S, Hashimoto M, Yoshiyama K, Kanemoto H, Hotta M, Azuma S, Suehiro T, Kakeda K, Nakatani Y, Umeda S, Fukuhara R, Takebayashi M, Ikeda M. Characteristics of behavioral symptoms in right-sided predominant semantic dementia and their impact on caregiver burden: a cross-sectional study. Alzheimers Res Ther. 2021 Oct 9;13(1):166. doi: 10.1186/s13195-021-00908-2. PMID 34627361

DOCUMENTS (1):
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT06218732/ICF_000.pdf